CLINICAL TRIAL: NCT07077655
Title: The Effectiveness of the Marmet Technique and Oxytocin Massage on Breast Milk Quantity in Mothers Who Have Undergone Cesarean Section
Brief Title: Marmet and Oxytocin Massage for Breast Milk Increase
Acronym: RCT
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Ege University (Other)
Responsible Party: Principal Investigator, Aysima Yalçıntepe, Midwife and Master's Student, Ege University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Other
Other Study IDs: EgeUniAYalc001
Record Dates: First submitted 2025-07-03; First posted 2025-07-22 (Actual); Last update posted 2025-09-22 (Actual); Status verified 2025-09

CONDITIONS: Healhty
Keywords: breastmilk; mother; massage techniques; marmet technique; oxytocin massage

STUDY DESIGN:
Intervention Model Description: In this study, there are three intervention groups. While two groups will receive an intervention, one group will serve as a placebo. The first group will be the Marmet technique group, the second group the oxytocin massage group, and the third group will be the placebo group. The study is designed as a randomized controlled single-blind study.
Who Masked: Participant
Masking Description: The study will be conducted in a single-blind design, meaning participants will be blinded to the intervention they receive. They will not be told what procedure is being performed; only the researcher will know.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- ARM1 (Marmet) (Active Comparator): One of the traditional and natural methods mothers can use to facilitate breast milk production after childbirth is the Marmet technique.
  Ensure hand hygiene and make sure the hands are warm. Ask the mother to remove her clothing/bra (assistance will be provided at this stage).
  Gently stroke the breast downward toward the nipple to trigger the let-down reflex.
  Starting from the armpit, move toward the breast, continuing the massage with circular finger movements around and toward the nipple.
  Ask the mother to lean forward slightly to allow gravity and gentle breast shaking to create mild vibrations and facilitate milk flow and drainage.
  After the procedure, assist the mother in adjusting her position assist the mother in adjusting her position and help her get dressed.
  Perform hand hygiene again. This procedure will be performed for 5 minutes on each breast, totaling 10 minutes, to ensure the technique is effective and standardized according to the literature.
  Interventions: Other: Marmet Technique
- ARM2 (Oxct.) (Active Comparator): Oxytocin massage is a technique applied to increase breast milk production. In this study, the following steps will be followed when performing oxytocin massage (Sari et al., 2017):
  Ensure hand hygiene and make sure the hands are warm. Ask the mother to remove her clothing/bra (assistance will be provided at this stage).
  Position the mother in a comfortable way (since all mothers in the oxytocin massage group will be within the first 2 hours post-cesarean, they will be positioned in bed, and if necessary, supported with pillows or rolled sheets).
  Using both thumbs facing forward, apply massage from the spine to the area beside the fifth and sixth ribs in a clockwise direction, first downward then upward.
  After the massage, gently wipe the mother's back with a paper towel (if she expresses discomfort).
  Assist the mother in adjusting her position and help her get dressed. Perform hand hygiene again. The massage will be applied for 3 minutes.
  Interventions: Other: Oxytocin Massage
- ARM3 (Plasebo) (Placebo Comparator): A light touch will be applied to the women's wrists, elbows, and shoulders.
  Interventions: Other: Plasebo

INTERVENTIONS:
Other: Marmet Technique — One of the traditional and natural efforts mothers can make to facilitate breast milk production postpartum is the Marmet technique. This technique embraces the principles of massage and stimulation of the milk ejection reflex (Widiastuti et al., 2015; Hairunisyah & Kusumawaty, 2022). Furthermore, this technique provides a relaxing effect, reactivating the milk ejection reflex, which in turn stimulates spontaneous milk flow (Yuliani et al., 2015). In other words, the Marmet technique is a combination of expressing milk and massaging the breast by emptying the lactiferous sinuses located under the areola. The Marmet technique stimulates prolactin secretion and helps maximize the milk ejection reflex. The more milk that is withdrawn or emptied from the breast, the greater the milk production (Widiastuti et al., 2015).
  Other Names: MarTec
  Arms: ARM1 (Marmet)
Other: Oxytocin Massage — Oxytocin massage is a type of massage performed to increase breast milk production. The massage is applied to the sides of the spine and the fifth to sixth ribs, and it stimulates the prolactin and oxytocin hormones after birth (Kosova et al., 2016). This massage serves to increase the oxytocin hormone, which can calm the mother, leading to an automatic flow of breast milk (Kilci & Sevil, 2021). Research conducted by Azizah and Ambarika (2022) shows that a combination of the Marmet technique and oxytocin massage can increase breast milk production. Massaging or stimulating the spine sends a message to the hypothalamus in the posterior pituitary by directly stimulating the medulla oblongata via neurotransmitters to release oxytocin, which then causes milk secretion from the breasts (Lestari & Linar, 2024).
  Other Names: OxyMas
  Arms: ARM2 (Oxct.)
Other: Plasebo — No intervention will be made to the participants in this group. Superficial touch will be performed on women's wrists, elbows, and shoulders.
  Arms: ARM3 (Plasebo)

SUMMARY:
This study is designed as a randomized controlled single-blind experimental study to examine the effectiveness of the oxytocin massage and Marmet technique applied to mothers who have undergone cesarean section on breast milk quantity and maternal state anxiety levels. The hypotheses of the study are as follows:

H0.1. There is no difference in the amount of breast milk among mothers in the Marmet technique, oxytocin massage, and control (placebo) groups.

H1.1. There is a difference in the amount of breast milk among mothers in the Marmet technique, oxytocin massage, and control (placebo) groups.

H0.2. There is no difference in the state anxiety scale scores among mothers in the Marmet technique, oxytocin massage, and control (placebo) groups.

H1.2. There is a difference in the state anxiety scale scores among mothers in the Marmet technique, oxytocin massage, and control (placebo) groups.

Participants:

Marmet technique, oxytocin massage, and control (placebo) groups will be informed about the study and asked to provide their consent. Participants will complete the descriptive questionnaire. Colostrum status will be checked and marked as "present" or "absent" on the "Breast Milk, Vital Signs, and Pain Level Form." Under researcher supervision, the mother will breastfeed her baby. Afterward, the State Anxiety Inventory will be administered.

Two hours later, mothers will express milk using a hospital-grade pump, with 15 minutes on each breast (total 30 minutes). Milk volume, vital signs, pain levels, and milk flow rate will be recorded on the relevant form. Following this, mothers in the Marmet group will receive 10 minutes of the Marmet technique, mothers in the oxytocin group will receive 5 minutes of oxytocin massage, and mothers in the control group will receive 5 minutes of light touch on their wrists and shoulders. Immediately after, milk expression will again be performed with 15 minutes per breast (30 minutes total). The State Anxiety Inventory will be re-administered, and milk amount, vital signs, pain levels, and flow rate will be recorded again.

All mothers will express milk using a hospital-grade breast pump, and the expression duration is standardized as 15 minutes per breast (30 minutes total) based on the literature. Two expressions will be performed - one before and one immediately after the intervention. Expressed milk will not be discarded and will instead be used to feed the babies via spoon or syringe under the researcher's supervision.

DETAILED DESCRIPTION:
This randomized controlled, single-blind experimental study aims to explore the physiological and psychological outcomes of two non-pharmacological breast stimulation techniques-oxytocin massage and the Marmet technique-on mothers who have undergone cesarean delivery. Specifically, the study investigates their effects on breast milk volume and maternal state anxiety levels during the early postpartum period.

Breastfeeding challenges are more commonly observed following cesarean deliveries due to delayed lactogenesis II, postoperative pain, mother-infant separation, and increased maternal stress. Non-invasive breast stimulation methods, such as the Marmet technique (which includes a structured pattern of massage, compression, and milk expression by hand) and oxytocin massage (which involves light tactile stimulation of the upper back and shoulders to promote oxytocin release), may provide physiological and psychological benefits to these mothers. This study systematically evaluates the efficacy of these techniques within a controlled hospital setting using standardized procedures.

Breast milk expression will be standardized using a hospital-grade electric pump, with a fixed pumping duration of 15 minutes per breast. Milk volume will be measured using calibrated collection containers provided with the pump. Vital signs (e.g., heart rate, blood pressure), self-reported pain levels (via Visual Analog Scale), and observed milk flow rate (rated as slow, moderate, or fast) will be recorded at each session.

Psychological impact will be assessed using the State-Trait Anxiety Inventory (STAI), focusing on the state anxiety subscale. This tool is a validated measure to assess transient anxiety responses under stress or in new environments, such as hospitalization or breastfeeding initiation after surgery.

The oxytocin massage protocol consists of light, rhythmic touch applied to the mother's upper arms, shoulders, and back for 5 minutes, aiming to stimulate endogenous oxytocin release through sensory nerve activation. The Marmet technique, applied for 10 minutes, follows a structured sequence of circular breast massage, downward milk movement, and manual expression techniques. The control group will receive light touch (5 minutes) applied to non-breast-related areas (wrists and shoulders) without known physiological effects on lactation or oxytocin release.

Post-intervention, mothers will perform a second round of milk expression under the same standardized conditions. Milk will not be discarded but will be fed to the infant using a spoon or syringe under researcher supervision, in accordance with neonatal nutrition safety standards.

This study is designed not only to measure lactation outcomes but also to consider maternal comfort and emotional state during the early postpartum phase, recognizing the interconnected nature of physiological milk production and maternal mental well-being. This study utilizes evidence-based lactation assessment methods and validated psychological scales. Data will be analyzed using IBM SPSS 20.0. Within-group and between-group comparisons will be conducted using paired t-tests and one-way ANOVA where appropriate. The study is approved by the relevant ethics committee and will adhere to Good Clinical Practice (GCP) guidelines.

ELIGIBILITY:
Inclusion Criteria:

* Aged between 18-35 years
* Literate
* Fluent in Turkish
* Volunteering to participate in the study
* Primiparous (first-time mothers)
* Within the first 2 hours postpartum (mothers performing their first breastfeeding under researcher supervision)
* Have a single baby with an appropriate birth weight for gestational age (>2500 gr)
* Have their baby with them
* Received spinal anesthesia
* Neither the mother nor the baby has any acute or chronic illness
* Exclusively breastfeeding their baby
* Had a term (37 weeks gestation or more) and cesarean delivery
* Experienced no complications after the cesarean section
* No issues preventing breastfeeding
* Willing to breastfeed

Exclusion Criteria:

* Are under 18 or over 35 years old
* Are multiparous (have given birth before)
* Are encountered more than 2 hours postpartum
* Received general anesthesia
* Have any acute or chronic illness themselves or their baby
* Have conditions requiring mother and baby to be separated
* Report experiencing severe pain
* Formula-feed their baby or consume any milk-increasing medication or tea
* Gave birth before 37 weeks gestation or had a vaginal delivery
* Have an anatomical breast issue (absence of nipple, inverted nipple)
* Have swelling, ecchymosis, or wounds on their back (for the oxytocin massage group)
* Have a baby with a congenital anomaly
* Have an issue preventing breastfeeding
* Have a psychological issue
* Are unwilling to breastfeed

Ages: 18 Years to 35 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Gender Based: Yes — Since only biological women produce breast milk, only women can participate in the study.
Enrollment: 123 (Estimated)
Dates: Start 2025-08-25 (Actual); Primary Completion 2025-12-30 (Estimated); Study Completion 2025-12-30 (Estimated)

PRIMARY OUTCOMES:
Breast milk volume | up to 4 months
  It's the amount of milk measured before and after the procedures applied to the mother.

SECONDARY OUTCOMES:
State Anxiety Scale Score | up to 4 months
  Participants' state anxiety levels will be measured before and after the intervention using the State Anxiety Scale. The minimum possible score on the State Anxiety Scale is 20, and the maximum is 80. Higher scores indicate higher levels of anxiety.

CONTACTS AND LOCATIONS:
Overall Officials: Aysima YALÇINTEPE, Principal Investigator — Ege University
Locations (1):
- Ege University Faculty of Medicine Hospital, Izmir, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Jutte J, Hohoff A, Sauerland C, Wiechmann D, Stamm T. In vivo assessment of number of milk duct orifices in lactating women and association with parameters in the mother and the infant. BMC Pregnancy Childbirth. 2014 Apr 2;14:124. doi: 10.1186/1471-2393-14-124. PMID 24694236
- [Background] Dhanawat A, Behura SS, Panda SK. Manual Method vs Breast Pump for Breast Milk Expression in Mothers of Preterm Babies During First Postnatal Week: A Randomized Controlled Trial. Indian Pediatr. 2022 Aug 15;59(8):608-612. doi: 10.1007/s13312-022-2572-8. PMID 35962654
- [Background] Zakarija-Grkovic I, Stewart F. Treatments for breast engorgement during lactation. Cochrane Database Syst Rev. 2020 Sep 18;9(9):CD006946. doi: 10.1002/14651858.CD006946.pub4. PMID 32944940
- [Background] Triansyah A, Stang, Indar, Indarty A, Tahir M, Sabir M, Nur R, Basir-Cyio M, Mahfudz, Anshary A, Rusydi M. The effect of oxytocin massage and breast care on the increased production of breast milk of breastfeeding mothers in the working area of the public health center of Lawanga of Poso District. Gac Sanit. 2021;35 Suppl 2:S168-S170. doi: 10.1016/j.gaceta.2021.10.017. PMID 34929803
- [Background] Alus Tokat M, Sercekus P, Yenal K, Okumus H. Early postpartum breast-feeding outcomes and breast-feeding self-efficacy in Turkish mothers undergoing vaginal birth or cesarean birth with different types of anesthesia. Int J Nurs Knowl. 2015 Apr;26(2):73-9. doi: 10.1111/2047-3095.12037. Epub 2014 Jun 5. PMID 24897921